CLINICAL TRIAL: NCT03087513
Title: Effect of Reversal of Neuromuscular Blockade on the Amplitude of Motor Evoked Potentials: A Randomized Controlled Crossover Study Comparing Sugammadex and Placebo
Brief Title: A Randomized Controlled Crossover Study Comparing Sugammadex and Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Associate Professor, Department of Anesthesia, Toronto Western Hospital, Toronto, Canada, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-5926-B
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Posterior Cervical Decompression and Fusion
Keywords: Motor Evoked Potentials, Spine surgery, Muscle relaxants
MeSH Terms: conditions — Muscle Hypotonia | interventions — Sugammadex; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized controlled crossover trial comparing the change in MEP amplitudes with administration of sugammadex or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized blinded study where the administering anesthetist, surgeon and neurophysiologists will be blinded to the intervention.
  Further, a blinded research assistant will perform assessment, data collection, and analysis of neurophysiology data attained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Initial Arm (Active Comparator): The study participants will receive either Sugammadex (2 mg/kg in 10 ml 0.9% normal saline) or placebo (10 ml of 0.9% normal saline).
  Interventions: Drug: Sugammadex Injection [Bridion]; Drug: Placebo
- Crossover Arm (Active Comparator): The study participants will receive the study medication that was not given in the initial arm (either Sugammadex (2 mg/kg in 10 ml 0.9% normal saline) or placebo (10 ml of 0.9% normal saline) .
  Interventions: Drug: Sugammadex Injection [Bridion]; Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex Injection [Bridion] — The study participants will receive 10 ml syringe containing Sugammadex (2mg/kg) in the first phase followed by Placebo 10 ml syringe containing of 0.9% of normal saline in the second phase.
  Other Names: Sugammadex
Drug: Placebo — The study participants will receive Placebo 10 ml syringe containing of 0.9% of normal saline in the first phase followed by 10 ml syringe containing Sugammadex (2mg/kg) in the second phase.
  Other Names: Normal Saline

SUMMARY:
Intraoperative monitoring of the motor evoked potentials has been shown to be both a sensitive and specific indicator for detecting intraoperative neurological injuries during spine surgery.(Fehlings, Brodke et al. 2010) It is utilized whenever there is risk for injury of nerve roots or the spinal cord during the procedure.

Anesthetic agents, especially the inhaled volatile anesthetics and muscle relaxants, are con-founders for motor evoked potential monitoring as they have deleterious effects on the amplitude of motor evoked potentials.(Sekimoto, Nishikawa et al. 2006) Hence, total intravenous anesthesia with no intraoperative muscle relaxants, are the standard anesthetic technique for these surgeries.

Muscle relaxants are usually required during the induction of anesthesia and endotracheal intubation of larynx. Current practice is to wait for the resolution of residual neuromuscular blockade before the motor evoked potential recordings (MEP) are initiated and this makes it difficult to assess if there was any neurological injury associated with positioning of the patient. A previous case series has shown that reversal of muscle relaxant can improve the amplitude of MEPs.(Batistaki, Papadopoulos et al. 2012) The aim of this study is to perform a randomized controlled trial to study the changes in motor evoked potential amplitudes comparing sugammadex and placebo.

DETAILED DESCRIPTION:
Motor evoked potential monitoring is a well-established and safe intervention to assist in prevention of intraoperative injury during spine surgery.(Schwartz, Sestokas et al. 2011) Patients with cervical myelopathy often present with neurological deficits and recording of the motor evoked potentials are often challenging in these patients. In addition, anesthetic agents especially muscle relaxants can abolish the motor response making it difficult to know when the baseline MEP can be recorded.

The usual anesthetic practice for patients undergoing posterior cervical spine surgery is to administer muscle relaxation to aid intubation at the start of the case . The neuromuscular blockade is then allowed to wear off and the neurophysiologist will attempt to record their baseline motor evoked potentials during or just prior to surgical exposure.

The issues with this current technique are;

1. Patients cannot be monitored for neurological changes during their transfer into the prone position
2. There is likely residual neuromuscular blockade decreasing the amplitude of motor evoked potentials.

Investigators plan to perform a randomized controlled cross-over trial comparing the change in MEP amplitudes with administration of sugammadex or placebo. This will be performed on at risk patients (e.g. cervical myelopathy) undergoing posterior cervical spine surgery where MEPs can be more difficult to attain but of higher utility.

The purpose of this study is to determine if reversal of residual neuromuscular blockade with Sugammadex can increase the amplitude of the motor evoked potentials.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18-80 years with American Society of Anesthesiologist (ASA) classification I-III undergoing cervical spine surgery in the prone position with intraoperative motor evoked potential monitoring.
* Operation time greater than 3 hours

Exclusion Criteria:

* Allergy to propofol or documented egg allergy
* Known allergy to sugammadex
* Severe renal dysfunction (EGFR<30)
* British Research Medical Council (BRMC) motor grading <3 in any peripheral muscle group preoperatively. This is inability to move the muscle group against gravity.
* Surgical requirement of strict muscle relaxation for surgical exposure
* Lack of informed consent
* Pregnancy
* Loss of MEP signals during washout period (or intraoperative spinal cord injury resulting in irreversible loss of MEP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, Principal Investigator — University Health Network, Toronto
Locations (1):
- TWH/UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venkatraghavan L, Royan N, Boyle SL, Dinsmore M, Lu N, Cushman K, Massicotte EM, Prabhu A. Effect of reversal of residual neuromuscular blockade on the amplitude of motor evoked potentials: a randomized controlled crossover study comparing sugammadex and placebo. Neurol Sci. 2022 Jan;43(1):615-623. doi: 10.1007/s10072-021-05318-8. Epub 2021 May 26. PMID 34041634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2018 and April 2019, 73 posterior cervical spine patients screened from the preoperative assessment clinic of Toronto Western Hospital to identify eligible patients.
  First participant was enrolled on March 2018 and the last participant was enrolled on April 2019.
Pre-assignment Details: 40 participants received 10ml syringe containing Sugammadex (2mg/kg) in the first phase, followed by Placebo 10 ml in the second phase or 10ml syringe containing Placebo in the first phase, followed by 10 ml of Sugammadex (2mg/kg) in the second phase.
  Time interval of approximately 3 hours between initial and crossover arm. 2 Patients withdrawn
Groups:
- Initial Arm and Crossover Arm: The study participants will receive either 10ml syringe containing Sugammadex (2mg/kg) or 10 ml Placebo 10 ml in the initial arm and in the crossover arm they will recieve the other drug ( sugammadex or Placebo) Washout period is 3 hours
Period: First Intervention
Arm/Group | Initial Arm and Crossover Arm
Started | 40
Completed | 40
Not Completed | 0
Period: Second Intervention After 3 hr Washout
Arm/Group | Initial Arm and Crossover Arm
Started | 40
Completed | 38
Not Completed | 2
Not completed — Equipment malfunction | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Intervention: Initial Arm The study participants will receive10ml syringe containing Sugammadex (2mg/kg) in the first phase, followed by 10 ml of Placebo in the second phase.
  Cross-over Arm The study participants will receive10ml syringe containing Placebo in the first phase, followed by 10 ml of Sugammadex (2mg/kg) in the second phase.
Arm/Group | Study Intervention
Number analyzed (Participants) | 38
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 60.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline Motor Evoked Potential amplitudes in both baseline and cross-over arms [Median (Inter-Quartile Range); unit: micro volts]
  Left FDI Sugammedex Group | 544.4 [165.8 to 1300]
  Left FDI Placebo Group | 377.1 [107.2 to 1650]
  Right FDI Sugammedex Group | 439.6 [101 to 1900]
  Right FDI Placebo Group | 418.7 [83.7 to 1425]

OUTCOME MEASURES:

1. Primary Outcome: Changes Motor Evoked Potentials (MEPs) Amplitude at 3 Minutes
Description: Changes in the amplitude of the Motor Evoked Potentials from the baseline in the first dorsal interosseous muscle at 3 minutes in sugammadex group compared to placebo group
Time Frame: Baseline and 3 minutes after the study intervention
Population: Data are presented as Median (IQR). MEP- Motor evoked potential, µV-microvolt, min-minute, 1Q- First quartile, 3Q-third quartile, FDI- first dorsal interosseous
Measure: Median (Inter-Quartile Range); unit: micro volts
Groups:
- Sugammadex: The study participants will receive a 10 ml syringe containing sugammadex (2mg/kg) in the first phase, followed by placebo 10 ml (0.9% normal saline) in the second phase.
- Placebo: The study participants will receive a 10ml syringe containing placebo (0.9% normal saline) in the first phase, followed by sugammadex 10 ml (2mg/kg) in the second phase.
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 38 | 38
micro volts
  Left FDI amplitude changes from baseline at 3 min | 652.9 [142 to 1650] | 20.6 [-183.5 to 297.5]
  Right FDI amplitude changes from baseline at 3 min | 2153.4 [1400 to 4536.8] | 55 [-65.2 to 480.8]
Statistical Analysis 1: Comparison: Sugammadex vs Placebo; In total, 40 patients were randomised for the study. Data from 2 patients were excluded as the crossover arm could not be completed due to intraoperative MEP change (n=1) and the equipment malfunction (n=1). The data distributions were tested for normality with the Kolmogorov-Smirnov test; Test type: Superiority; p < 0.01, Mixed Models Analysis — In all cases of motor evoked potential changes, a P-value of 0.05 was considered significant; As the amplitude values were non-normally distributed, the Mann-Whitney U test was performed to compare the two groups

2. Secondary Outcome: MEPs Amplitude Changes in Both Sugammadex and Placebo Groups
Description: Changes in the amplitude of the MEPs from the baseline in the first dorsal interosseous muscle at 6 minutes
Time Frame: Baseline to 6 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: micro volts
Groups:
- Sugammadex Group: The study participants will receive a 10ml syringe containing sugammadex (2mg/kg) in the first phase, followed by placebo (10 ml of 0.9% normal saline) in the second phase.
- Placebo Group: The study participants will receive a 10 ml syringe containing placebo (0.9% normal saline) in the first phase, followed by sugammadex 10 ml (2mg/kg) in the second phase.
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 38 | 38
micro volts
  Left FDI | 646.4 [253.1 to 1580.9] | 84.3 [-178.6 to 679.8]
  Right FDI | 1609.3 [632.4 to 5535.7] | 201.9 [-0.525 to 760.7]

3. Secondary Outcome: MEPs Amplitude Changes From Baseline at 9 Minutes
Description: Comparison of changes in MEP amplitudes from baseline at 9 minutes between sugammadex and placebo groups
Time Frame: Baseline to 9 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: micro volts
Groups:
- Sugammedex Group: The study participants will receive a 10ml syringe containing sugammadex (2mg/kg) in the first phase, followed by placebo (10 ml 0.9% normal saline) in the second phase.
Arm/Group | Sugammedex Group | Placebo Group
Number analyzed (Participants) | 38 | 38
micro volts
  Left FDI | 894.9 [234.1 to 2261.2] | 105.5 [-115.2 to 775]
  Right FDI | 1256.3 [308.9 to 2533.1] | 337.2 [-17.5 to 2215.8]

4. Secondary Outcome: Patient Movement
Description: Number of patients moved and observed by the surgeon. From the study intervention to the surgeon observed patient movements
Time Frame: From 0 to 15 minutes
Measure: Number; unit: participants
Groups:
- Sugammadex Group: The study participants will receive a 10ml syringe containing sugammadex (2mg/kg) in the first phase, followed by placebo (10 ml 0.9% normal saline) in the second phase.
- Placebo Group: The study participants will receive a 10ml syringe containing placebo (0.9% normal saline) in the first phase, followed by sugammadex 10 ml (2mg/kg) in the second phase.
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 38 | 38
participants | 6 | 0

5. Secondary Outcome: Surgical Grading of Relaxation of the Surgical Field
Description: Surgical grading of relaxation of the surgical field as per the Likert-4 point surgical grading of surgical field.
  During surgical exposure and closure.
Time Frame: approximatelt 1 hour - 30 min during surgical exposure and 30 minutes during closure
Measure: Count of Participants; unit: Participants
Groups:
- Sugammadex: The study participants will receive a 10ml syringe containing sugammadex (2mg/kg) in the first phase, followed by placebo 10 ml in the second phase.
- Placebo: The study participants will receive a 10ml syringe containing placebo in the first phase, followed by sugammadex 10 ml (2mg/kg) in the second phase.
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 38 | 38
Participants
  Good or optimal condition | 31 | 35
  Acceptable | 6 | 3
  Poor | 1 | 0

ADVERSE EVENTS:
Time Frame: From the study intervention to the end of surgery, approximately 3 hours
Description: All adverse events occurring during the study intervention period.
Arm/Group | Sugammadex Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03087513/Prot_SAP_000.pdf